CLINICAL TRIAL: NCT04533776
Title: Peer-Interaction Group Support in Adolescents With Celiac Disease: A Randomized Controlled Trial
Brief Title: Support for Adolescents With Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melike Taşdelen Baş (Other)
Responsible Party: Sponsor-Investigator, Melike Taşdelen Baş, Lecturer, Dr.(Nursing Department), Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/08-24 (KA-180047)
Record Dates: First submitted 2020-08-10; First posted 2020-09-01 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Celiac Disease in Children
Keywords: Celiac Disease; Adolescent; Quality of Life; Friendship Relations; Coping; Nursing Care
MeSH Terms: conditions — Celiac Disease | interventions — Therapeutics; Diet, Gluten-Free; Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEER-INTERACTION GROUP SUPPORT (Experimental): All the sessions of the research took place in a classroom in the hospital. The sessions lasted an average of 90 minutes with two 45-minute sections. During the break, which lasted about 20 minutes, gluten-free products were offered. During the break, adolescents were given the opportunity to chat and interact with each other.
  Peer interactive group support was implemented for 3 months with an interval of one week. A total of 6 sessions were held with the study group. Adolescents in the study group were contacted by phone before each session. The day before the session, a text message was sent to all participants informing the location and time of the meeting. The contents of the first and second sessions in relation to the study were created beforehand. However, contents of the third, fourth, fifth and sixth sessions were prepared after the first two sessions.
  Interventions: Behavioral: Celiac Disease Definition, Symptoms and Treatment; Behavioral: Difficulties Due to Celiac Disease; Behavioral: Gluten Free Diet in Celiac Disease; Behavioral: Difficulties Related to Disease in School and Social Life; Behavioral: Celiac Disease and Its Effects on Acamdemic Success Peer Relations; Behavioral: Celiac Diseae anf Future Goals
- routine health care- control group (Experimental): Peer interactive group support was not provided to the control group.
  Interventions: Other: No Intervention: routine health care- control group

INTERVENTIONS:
Behavioral: Celiac Disease Definition, Symptoms and Treatment — * Adolescents share their knowledge about the disease
  * Emphasizing the definition and symptoms of celiac disease
  * Discussion of the treatment of celıac disease Expression Question-Answer Discussion Summarizing
  Arms: PEER-INTERACTION GROUP SUPPORT
Behavioral: Difficulties Due to Celiac Disease — * Determining what experience living with celiac is fot the patient (What do I think about the disease, how do I feel about the disease,how do I perceive the disease, how does the disease affect me)
  * Determining the difficulties encountered in Daily life due to illness (How do I deal with difficulties)
  * Determining how the disease affects life Expression Question-Answer Discussion Summarizing
  Arms: PEER-INTERACTION GROUP SUPPORT
Behavioral: Gluten Free Diet in Celiac Disease — * Evaluating dietary information
  * Identifying the difficulties in diet therapy Expression Question-Answer Discussion Summarizing Case Study Presentation (Transfer of life experience of an individual who is 22 years old with celiac disease)
  Arms: PEER-INTERACTION GROUP SUPPORT
Behavioral: Difficulties Related to Disease in School and Social Life — * Assessment of difficulties encountered in school and social life
  * Evaluation of the solution suggestions fort he difficulties encountered Expression Question-Answer Discussion Summarizing Örnek Olay Sunumu (Transfer of life of experience of a 23 years old dietician with celiac disease)
  Arms: PEER-INTERACTION GROUP SUPPORT
Behavioral: Celiac Disease and Its Effects on Acamdemic Success Peer Relations — * Evaluation of the effects of the disease on academic success
  * Evaluation of the effects of the disease on peer relationships in the school enviroment
  * Difficulties experienced in peer relations and evaluation of relationships (exclusion) Expression Question-Answer Discussion Summarizing
  Arms: PEER-INTERACTION GROUP SUPPORT
Behavioral: Celiac Diseae anf Future Goals — * General summary of all sessions so far
  * Summarizing the topics discussed in the previous session
  * Evaluating the future goals of the participants Expression Question-Answer Discussion Summarizing
  Arms: PEER-INTERACTION GROUP SUPPORT
Other: No Intervention: routine health care- control group — Peer interactive group support was not provided to the control group. After all the sessions of the peer interactive group support of the study were completed, a separate training meeting was held for the control group.
  Arms: routine health care- control group

SUMMARY:
This study was designed as a randomized controlled experimental study to examine the effects of peer-interaction group support in adolescents with celiac disease (CD) in the 13-18 age group on the quality of life, friendship relations, and coping levels of adolescents.

Six peer interactive group sessions were held with one week intervals with adolescents (n = 18) in the study group included in the sample for a period of 3 months. In the sessions, all participants were asked questions about the purpose of the session and a discussion environment was created. No training and counseling were provided to the adolescents in the control group (n = 18). Before and after the peer interactive group support, adolescents in the intervention and control group were asked to complete the quality of life, friendship qualities, and coping scales.

DETAILED DESCRIPTION:
The study is a randomized controlled experimental study conducted to examine the effect of peer interactive group support on quality of life, peer relationships and coping (coping) levels in adolescents aged 13-18 years with celiac disease.

The study was conducted on adolescents with a diagnosis of celiac disease in the outpatient clinic of the Department of Child Health of Afyon Kocatepe University in Afyonkarahisar. This change took place after research permissions were obtained. Patients are served in the polyclinic between 09:00 and 17:00 on weekdays. Gastroenterology Specialist, who monitors the patients with Celiac diagnosis, works as a physician. There are no nurses in the polyclinic and individual training is not given to celiac patients according to their needs.

There are 85 patients with a diagnosis of celiac disease in the 0-18 age group who were followed up in the Department of Child Health and Diseases of Afyonkarahisar Health Sciences University, where the study will be conducted. It was determined from the patient records that there were 36 patients with a diagnosis of celiac disease in the 13-18 age group. The universe of the study consisted of patients with a diagnosis of celiac disease in the 13-18 age group who were followed up in the Pediatric Outpatient Clinic of Afyonkarahisar University of Health Sciences.

Data Collection Tools Introductory Information Form, Quality of Life Scale for Children (13-18 age group), Friendship Qualities Scale and Coping Scale for Adolescents prepared by the researcher for data collection.

Introductory Information Form In this form prepared by the researcher, there are 14 questions regarding the demographic characteristics of the mother, father, family and child. After randomization, an introductory information form (before peer interactive group support) was administered to all adolescents in the research and control groups in a classroom of the Pediatric Outpatient Clinic where the study was conducted.

Children's Quality of Life Scale - PedsQL (13-18 age group) The quality of life scale for children was developed by Varni et al. (1999) to measure the quality of life of children and adolescents aged 2-18 years. The internal consistency coefficient (Cronbach's alpha) of the section prepared for children of the scale developed by Varni et al. Was found to be 0.93. Memik et al. (2007) conducted a study on the validity and reliability of the adolescent form of the PedsQL (13-18 years old).

While the World Health Organization defines health, it covers the areas of physical, emotional and social functionality. Scoring is made for these three areas in the scale. In the scale, a fourth area under the name of school functionality is questioned. The psychosocial health total score (PSTP) is calculated by calculating the total score (STP), physical health total score (FSTP), emotional, social and school functionality item scores in the scale.

The Quality of Life Scale for Children (PedsQL) is a scale suitable for use in healthy or ill children and adolescents in settings such as schools and hospitals. The scale consists of 23 items in total. The scale is in the form of a 5-point Likert scale and is scored between 0-4. The items are scored between 0-100. The scale gives 100 points for never answer, rarely 75 points for its answer, sometimes 50 points for its answer, often 25 points for its answer, and almost always 0 points for its answer. The Turkish validity and reliability study of the PedsQL for the 13-18 age group was conducted by Memik et al. (2007). The internal consistency coefficient (Cronbach's alpha) of the form prepared for adolescents in the study of Memik et al. Was found to be 0.82.

Friendship Qualities Scale The friendship qualities scale aims to evaluate the relationships of 10-18 year old children and adolescents with their best friends. The scale was created by Bukowski et al. (1994). The internal consistency coefficients (Cronbach's alpha) according to the sub-dimensions of the scale were: 0.72; conflict: 0.68; proximity: 0.76; help: 0.81; and protection: found to be 0.58. The Turkish validity and reliability study of the scale was conducted by Erkan Atik et al. (2014). Participants included in the study are secondary and high school students. The internal consistency coefficient of the whole scale in the study of Erkan Atik et al. Was found to be 0.85. The scale includes 22 items and five sub-dimensions. The scale is graded from 1 to 5. "1" is not right for your friendship, "2" may be correct, "3" is usually correct, "4" is very correct, "5" is completely correct. The sub-dimensions of the scale are togetherness, conflict, assistance, protection and closeness. Togetherness sub-dimension, items 1, 2, 3 and 4, conflict sub-dimension 5,6,7 and 8 items, help sub-dimension 9,10,11,12 and 13 items, protection sub-dimension 14,15,16 and 17th items, proximity sub-dimension is calculated by evaluating items 18,19,20,21 and 22. All items in the conflict sub-dimension of the scale are calculated by reverse coding. The scores that can be obtained vary between 4-20 in the Togetherness, Conflict and Protection sub-dimensions, and 5-25 in the Assistance and Proximity sub-dimensions. If the scale score to be obtained from both the total score and the sub-dimensions is high, this is considered as positive peer relationships.

Coping Scale for Adolescents (KIDCOPE) The scale, which was created by Spirito et al. (1988) under the name of KIDCOPE (multidimensional coping strategies for children scale), consists of two forms for children (5-13 years old) and adolescents (13-18 years). The internal consistency coefficient (Cronbach's alpha) of the scale was 0.62. The Coping Scale for Adolescents consists of 11 items in total. This scale includes ten coping strategies. These strategies include social distancing, distraction, desiring thinking, problem solving, withdrawal, cognitive restructuring, social support, emotion regulation, self-criticism, and blaming others.

The 10 strategies included in KIDCOPE are; distraction (played a game to watch or forget TV), withdrawal (left alone), desiresing thinking (wanted to be able to do things differently), self-criticism (blamed myself), blaming others (blaming someone else for causing the problem), problem solving (I tried to solve the problem by thinking about the answers), emotion regulation (tried to calm myself or yelled, screamed), cognitive restructuring (tried to see the good side of things), social support (tried to feel better by spending time with family or friends) and social distancing (I didn't want to spend time with my family or friends) The 10 strategies included in KIDCOPE are; distraction (played a game to watch or forget TV), withdrawal (left alone), desiresing thinking (wanted to be able to do things differently), self-criticism (blamed myself), blaming others (blaming someone else for causing the problem), problem solving (I tried to solve the problem by thinking about the answers), emotion regulation (tried to calm myself or yelled, screamed), cognitive restructuring (tried to see the good side of things), social support (tried to feel better by spending time with family or friends) and social distancing (I didn't want to spend time with my family or friends) In the implementation phase of the study, a classroom belonging to the Child Health and Diseases Polyclinic of Afyonkarahisar Health Sciences University Faculty of Medicine Hospital was used. All sessions in the research were held in this classroom. The sessions lasted an average of 90 minutes in two 45-minute sections. Gluten-free products were presented during the 20-minute break between sessions. During the break, adolescents were given the opportunity to interact with each other by chatting. The pre-test application of the introductory information form and scale forms of all the participants in the research group was applied at the beginning of the first session, and the post-test application at the end of the last session, which was the sixth session. The pre-test application of the participants included in the control group was applied on the same day separately from the research group, and the post-test application (only scales) was applied in the same classroom at the end of all sessions.

Research Group Interactive peer group support was implemented for 3 months, one week apart. A total of 6 sessions were held with the research group. Group meetings were planned to be held at the weekend in order to prevent adolescents' attendance at school. However, as the data collection phase is in the summer and schools are closed, the sessions were held on weekdays and bi-weekly. The adolescents in the study group were reached by phone before each session. One day before the session, all participants were sent a text message informing the meeting and its place and time and they were invited. Each session lasted 1.5 hours on average.

The contents of the first and second sessions of the research were prepared beforehand. However, the contents of the third, fourth, fifth and sixth sessions were arranged after the first two sessions. Table of contents of the 6 sessions held is presented in Table 3.

In the sessions, all participants were asked questions regarding the target determined for the session. By creating a discussion environment based on these questions, it was ensured that the participants shared their problems and solutions with each other. The responses of the participants to the questions were noted and reported by the researcher.

Control Group No peer interactive group support was provided to the control group. In the control group, in a classroom belonging to the University's Child Health and Diseases Polyclinic where the study was conducted, the Introductory Information Form, the Quality of Life Scale for Children, the Friendship Qualities Scale, the Adolescent Coping Scale were applied after the adolescents and parents were informed about the subject of the study and written permission was obtained. Three months later, the Adolescents in the control group were administered the Quality of Life Scale for Children, Friendship Qualities Scalee, and the Adolescent Coping Scale.

The adolescents in the control group were not informed about the routine education they received from the hospital during the study. A separate training meeting was held for the control group on 11.10.2018, after all sessions of the peer interactive group support of the study were completed. The training lasted about one hour in the classroom of the University's Child Health and Diseases Polyclinic. The definition, symptoms and signs of celiac disease, treatment and dietary rules were discussed in the training content. At the end of the meeting, an information booklet titled "Living with Celiacs" was given.

ELIGIBILITY:
Inclusion Criteria:

* Must have had celiac disease for more than a year
* Must be between 13-18 years old

Exclusion Criteria:

* Another chronic disease
* Psychiatric illness

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life Scale | 12 weeks
  The Quality of Life Scale for Children (PedsQL) is a scale suitable for use in healthy or ill children and adolescents in settings such as schools and hospitals. The scale consists of 23 items in total. The scale is in the form of a 5-point Likert scale and is scored between 0-4. The items are scored between 0-100. It is thought that the higher the total score for PedsQL, the better the health-related quality of life.
Friendship Qualities Scale | 12 weeks
  Friendship Qualities Scale The Friendship Qualities Scale aims to evaluate the relationship of children and adolescents in the 10-18 age group with their best friends. The scores that can be obtained vary between 4-20 in the Togetherness, Conflict and Protection sub-dimensions, and 5-25 in the Assistance and Proximity sub-dimensions. If the scale score to be obtained from both the total score and the sub-dimensions is high, this is considered as positive peer relationships.
Coping Scale (KIDCOPE) | 12 weeks
  Coping Scale for Adolescents (KIDCOPE) The scale, which was created by Spirito et al. (1988) under the name of KIDCOPE (multidimensional coping strategies for children scale), consists of two forms for children (5-13 years old) and adolescents (13-18 years).The scores to be scored range from 0-12 for active and avoidant coping, and 0-9 points for negative coping. A higher score indicates that the assessed coping approach is used more.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Çavuşoğlu, Study Director — Hacettepe University
Locations (1):
- Selcuk University Aksehir Kadir Yallagöz Health School., Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-sheyab N, Gallagher R, Crisp J, Shah S. Peer-led education for adolescents with asthma in Jordan: a cluster-randomized controlled trial. Pediatrics. 2012 Jan;129(1):e106-12. doi: 10.1542/peds.2011-0346. Epub 2011 Dec 12. PMID 22157137
- [Background] de Lorenzo CM, Xikota JC, Wayhs MC, Nassar SM, de Souza Pires MM. Evaluation of the quality of life of children with celiac disease and their parents: a case-control study. Qual Life Res. 2012 Feb;21(1):77-85. doi: 10.1007/s11136-011-9930-7. Epub 2011 May 20. PMID 21598063
- [Background] Errichiello S, Esposito O, Di Mase R, Camarca ME, Natale C, Limongelli MG, Marano C, Coruzzo A, Lombardo M, Strisciuglio P, Greco L. Celiac disease: predictors of compliance with a gluten-free diet in adolescents and young adults. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):54-60. doi: 10.1097/MPG.0b013e31819de82a. PMID 19644397
- [Background] Fasano A, Catassi C. Clinical practice. Celiac disease. N Engl J Med. 2012 Dec 20;367(25):2419-26. doi: 10.1056/NEJMcp1113994. No abstract available. PMID 23252527
- [Background] Hill ID, Dirks MH, Liptak GS, Colletti RB, Fasano A, Guandalini S, Hoffenberg EJ, Horvath K, Murray JA, Pivor M, Seidman EG; North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. Guideline for the diagnosis and treatment of celiac disease in children: recommendations of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. J Pediatr Gastroenterol Nutr. 2005 Jan;40(1):1-19. doi: 10.1097/00005176-200501000-00001. PMID 15625418
- [Background] Kautto E, Ryden PJ, Ivarsson A, Olsson C, Norstrom F, Hogberg L, Carlsson A, Hagfors L, Hornell A. What happens to food choices when a gluten-free diet is required? A prospective longitudinal population-based study among Swedish adolescent with coeliac disease and their peers. J Nutr Sci. 2014 Feb 13;3:e2. doi: 10.1017/jns.2013.24. eCollection 2014. PMID 25191610
- [Background] Lebwohl B, Sanders DS, Green PHR. Coeliac disease. Lancet. 2018 Jan 6;391(10115):70-81. doi: 10.1016/S0140-6736(17)31796-8. Epub 2017 Jul 28. PMID 28760445
- [Background] Newton KP, Singer SA. Celiac disease in children and adolescents: special considerations. Semin Immunopathol. 2012 Jul;34(4):479-96. doi: 10.1007/s00281-012-0313-0. Epub 2012 May 2. PMID 22549889
- [Background] Rose C, Howard R. Living with coeliac disease: a grounded theory study. J Hum Nutr Diet. 2014 Feb;27(1):30-40. doi: 10.1111/jhn.12062. Epub 2013 Mar 21. PMID 23516989
- [Background] Sevinc E, Cetin FH, Coskun BD. Psychopathology, quality of life, and related factors in children with celiac disease. J Pediatr (Rio J). 2017 May-Jun;93(3):267-273. doi: 10.1016/j.jped.2016.06.012. Epub 2016 Nov 23. PMID 27886806
- [Result] Biagetti C, Naspi G, Catassi C. Health-related quality of life in children with celiac disease: a study based on the Critical Incident Technique. Nutrients. 2013 Nov 12;5(11):4476-85. doi: 10.3390/nu5114476. PMID 24225846
- [Result] Bongiovanni TR, Clark AL, Garnett EA, Wojcicki JM, Heyman MB. Impact of gluten-free camp on quality of life of children and adolescents with celiac disease. Pediatrics. 2010 Mar;125(3):e525-9. doi: 10.1542/peds.2009-1862. Epub 2010 Feb 15. PMID 20156892
- [Result] Cai RA, Holt RIG, Casdagli L, Viner RM, Thompson R, Barnard K, Christie D. Development of an acceptable and feasible self-management group for children, young people and families living with Type 1 diabetes. Diabet Med. 2017 Jun;34(6):813-820. doi: 10.1111/dme.13341. PMID 28226183
- [Result] Chauhan JC, Kumar P, Dutta AK, Basu S, Kumar A. Assessment of dietary compliance to gluten free diet and psychosocial problems in Indian children with celiac disease. Indian J Pediatr. 2010 Jun;77(6):649-54. doi: 10.1007/s12098-010-0092-3. Epub 2010 Jun 8. PMID 20532683
- [Result] Creedy D, Collis D, Ludlow T, Cosgrove S, Houston K, Irvine D, Fraser J, Moloney S. Development and evaluation of an intensive intervention program for children with a chronic health condition: a pilot study. Contemp Nurse. 2004 Dec-2005 Jan;18(1-2):46-56. doi: 10.5172/conu.18.1-2.46. PMID 15729797
- [Result] Eisenberg SA, Shen BJ, Schwarz ER, Mallon S. Avoidant coping moderates the association between anxiety and patient-rated physical functioning in heart failure patients. J Behav Med. 2012 Jun;35(3):253-61. doi: 10.1007/s10865-011-9358-0. Epub 2011 Jun 10. PMID 21660588
- [Result] Jaser SS, White LE. Coping and resilience in adolescents with type 1 diabetes. Child Care Health Dev. 2011 May;37(3):335-42. doi: 10.1111/j.1365-2214.2010.01184.x. Epub 2010 Dec 9. PMID 21143270
- [Result] Klein DM, Turvey CL, Pies CJ. Relationship of coping styles with quality of life and depressive symptoms in older heart failure patients. J Aging Health. 2007 Feb;19(1):22-38. doi: 10.1177/0898264306296398. PMID 17215200
- [Result] Kolsteren MM, Koopman HM, Schalekamp G, Mearin ML. Health-related quality of life in children with celiac disease. J Pediatr. 2001 Apr;138(4):593-5. doi: 10.1067/mpd.2001.111504. PMID 11295729
- [Result] Mackner LM, Ruff JM, Vannatta K. Focus groups for developing a peer mentoring program to improve self-management in pediatric inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2014 Oct;59(4):487-92. doi: 10.1097/MPG.0000000000000473. PMID 24979662
- [Result] Scheel A, Beaton A, Okello E, Longenecker CT, Otim IO, Lwabi P, Sable C, Webel AR, Aliku T. The impact of a peer support group for children with rheumatic heart disease in Uganda. Patient Educ Couns. 2018 Jan;101(1):119-123. doi: 10.1016/j.pec.2017.07.006. Epub 2017 Jul 11. PMID 28716486
- [Result] Smeulders ES, van Haastregt JC, Ambergen T, Uszko-Lencer NH, Janssen-Boyne JJ, Gorgels AP, Stoffers HE, Lodewijks-van der Bolt CL, van Eijk JT, Kempen GI. Nurse-led self-management group programme for patients with congestive heart failure: randomized controlled trial. J Adv Nurs. 2010 Jul;66(7):1487-99. doi: 10.1111/j.1365-2648.2010.05318.x. Epub 2010 May 21. PMID 20492026
- [Result] Snead K, Ackerson J, Bailey K, Schmitt MM, Madan-Swain A, Martin RC. Taking charge of epilepsy: the development of a structured psychoeducational group intervention for adolescents with epilepsy and their parents. Epilepsy Behav. 2004 Aug;5(4):547-56. doi: 10.1016/j.yebeh.2004.04.012. PMID 15256193
- [Result] Stewart M, Letourneau N, Masuda JR, Anderson S, McGhan S. Impacts of online peer support for children with asthma and allergies: It just helps you every time you can't breathe well". J Pediatr Nurs. 2013 Sep-Oct;28(5):439-52. doi: 10.1016/j.pedn.2013.01.003. Epub 2013 Feb 9. PMID 23398896
- [Result] Trivedi RB, Blumenthal JA, O'Connor C, Adams K, Hinderliter A, Dupree C, Johnson K, Sherwood A. Coping styles in heart failure patients with depressive symptoms. J Psychosom Res. 2009 Oct;67(4):339-46. doi: 10.1016/j.jpsychores.2009.05.014. PMID 19773027

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT04533776/Prot_SAP_ICF_000.pdf